CLINICAL TRIAL: NCT00273676
Title: Costs and Effects of Early Switch of Intravenous to Oral Antibiotics in Severe Community-Acquired Pneumonia: a Multicenter Randomized Trial
Brief Title: Study on Costs and Safety of Early Conversion From Intravenous to Oral Antibiotic Treatment in Patients With Severe Community-Acquired Pneumonia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Dutch Health Care Insurance Board (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OG 99-64
Record Dates: First submitted 2006-01-05; First posted 2006-01-09 (Estimated); Last update posted 2006-01-09 (Estimated); Status verified 2006-01

CONDITIONS: Severe Communtity-Acquired Pneumonia
Keywords: Community-acquired pneumonia; Treatment; Antibiotics
MeSH Terms: conditions — Community-Acquired Pneumonia

INTERVENTIONS:
Procedure: Conversion to oral antibiotic treatment after 3 days of intravenous antibiotic treatment

SUMMARY:
Patients with severe community-acquired pneumonia are included Half of the patients are treated with a 3 day course of intravenous antibiotics, followed, when clinical stable, by a course of oral antibiotics. Efficacy of this treatment is compared to a standard course of 7 days of intravenous antibiotics, which treatment is assigned to the other half of patients. Outcomes measured are clinical cure and costs.

DETAILED DESCRIPTION:
Study design A multi-center, randomized open label clinical trial was performed in 2 university medical centers and 5 teaching hospitals in the Netherlands. The study was approved by the medical ethics committees of all participating hospitals and all patients provided written informed consent prior to enrollment.

After inclusion in the trial, treatment allocation was established through an independent central randomization center. Stratified randomization per center was based on computer generated tables. Patients were either randomized to the intervention group, where clinically stable patients were switched from IV to oral antibiotics on the 3rd day of hospitalization to complete a total of 10 days antibiotic treatment, or to the control group, who received a standard regimen of 7 days of intravenous therapy. Clinical stability was defined as respiratory rate < 25/min, O2 saturation > 90% or arterial pO2>55mmHg, hemodynamically stable, > 1oC decrease in temperature in case of fever, absent mental confusion and the ability to take oral medication 10. Antibiotic choices were left to the discretion of the attending consultant and were based on Dutch treatment guidelines 20.

Patients Adult patients (age 18 or above) with severe CAP admitted to general hospital wards were eligible for inclusion in the study. Pneumonia was defined as a new or progressive infiltrate on a chest X-ray plus at least two of the following criteria: cough, sputum production, rectal temperature > 38oC or < 36.1oC, auscultatory findings consistent with pneumonia, leucocytosis (>10.000/mm3, or >15% bands), C-reactive protein > 3 times the upper limit of normal, positive blood culture or positive culture of pleural fluid. 21 Severe pneumonia was defined as Fine class IV or V or fulfilling the ATS-criteria for severe community-acquired pneumonia. 16;22 Patients with cystic fibrosis, a history of colonization with Gram negative bacteria due to structural damage to the respiratory tract, malfunction of the digestive tract, life expectancy of less than 1 month due to underlying diseases, infections other than pneumonia needing antibiotic treatment, severe immunosuppression (neutropenia (<0,5 x 109 / l) or a CD4 count < 200 / mm3) and needing mechanical ventilation in an intensive care unit were excluded.

Baseline, follow up and outcome measurements Patients were followed for a maximum of 28 days. On admission, a complete physical examination, chest radiography and blood sampling for arterial blood gas analysis and for hematological and biochemical analysis were performed. Demographic data, initial intravenous therapy and clinical data were recorded. During the follow-up period, in-hospital clinical data were recorded. Clinical stability was evaluated after 3 days of intravenous therapy in both study groups and discharge criteria (temperature < 37.8 oC, saturation >92%, normal blood pressure, heart rate < 100/min, respiratory rate < 25/min, absence of mental confusion and ability to take oral medication ) were evaluated daily thereafter. If patients were discharged within 28 days after admission they were asked to return to the out-patient clinic 28 days after inclusion, where history, physical examination, blood chemistry analysis and a chest X-ray were taken and health-care consumption after discharge was recorded.

Questionnaires were used to evaluate the effects on health care resource use outside the hospital (recorded daily after discharge). Quality of life was determined with the short form health survey questionnaire (www.sf-36.org) recorded at days 3, 10 and 28 of the study. Additional questionnaires were used to measure the effects of an early discharge on the workload for family members (questionnaire at day 28 of study) and effects of administration route on freedom of movement, adverse events and compliance (questionnaire at day 7 of study). Treatment failures were defined as death, clinical deterioration (clinical worsening such that the patient needed mechanical ventilation, re-administration of intravenous antibiotics after a switch to oral therapy, readmission for pulmonary reinfection after discharge, increase in temperature after initial improvement) or hospitalization at day 28 of the study. Clinical cure was defined as discharged in good health without signs and symptoms of pneumonia and no treatment failures during the follow-up period. 21

Microbiological analyses Sputum samples and blood samples were collected, cultured and evaluated following standard procedures. Micro-organisms cultured in blood or sputum were recorded. In addition, Binax NOW-tests were used to detect urinary antigen for Legionella pneumophila and S. pneumoniae. Acute and convalescent serology samples were collected and evaluated for Mycoplasma pneumoniae, L. pneumophila and Chlamydia pneumonia. Any non-contaminating micro-organism cultured from a blood or sputum sample or detected by urinary antigen testing was considered a cause for the episode of pneumonia. For Mycoplasma pneumoniae, a fourfold or greater increase in titer in paired sera or a single titer of greater than or equal to 1:40 was considered indicative of infection. 23 (Immune fluorescence agglutination, Serodia-MycoII ®, Fujirebio, inc.) For Legionella pneumophila, a fourfold increase in the antibody titer to 1:128 or greater, or single titers of 1:256 or more were considered suggestive of Legionella pneumonia.24 For Chlamydia pneumoniae, detection of IgM above established values, seroconversion of IgG between acute and convalescence samples, high amounts of IgG in single titers or a combination of these factors were considered serological evidence of infection, according to the manufacturers instructions. (ELISA, Savyon Diagnostics Ltd)

Economic evaluation The societal perspective was used to calculate direct medical costs associated with the treatment in both study groups. Costs were assessed in 2002 euros. Costs per patient were calculated by multiplying resource use by the unit costs. Resource use during hospital stay for diagnostic and therapeutic interventions, consultations of medical or paramedic specialists and antibiotic use was measured. Resource use outside the hospital was evaluated using questionnaires which recorded contacts with general practitioners, specialists, extra diagnostic procedures, use of medication, readmissions, home care and other disease-related costs. Additional costs associated with specific diagnostic tests were based on tariffs. Costs of hospital stay, diagnostic procedures and specialist consultations, were calculated using unit costs as determined within the realm of the Dutch guidelines for pharmaco-economic analyses 25. Costs for readmissions and reinfections were assessed specifically for the study cohort and included costs for extra diagnostic procedures, treatment and hospitalizations. Costs of antibiotics prescribed were estimated using Dutch 2002 formulary cost-prices 26

Sample size and statistical analysis To demonstrate equivalence in efficacy of the two treatment groups, initially, the sample size was set at 250 patients in each study group based on an expected cure rate of 85% in the IV group and acceptance of a 75% cure rate in the switch group. (=0.05, 2 sided; 1-=0.80). The absolute difference in cure rate including 95% CI was calculated. Equivalence was rejected if the lower limit of the CI exceeded -10%. Eventually, with less than anticipated enrolment, a 15% lower effectiveness in the intervention group could be excluded with =0.05 and 1-=0.80.

Analyses were performed on an intention-to-treat basis. Differences in continuous variables were presented as absolute differences with their corresponding 95% CI´s. Dichotomous data were compared with chi-square statistics. Alike cure rate differences in proportions were presented including 95% CI´s. For cost-calculations, arithmetic means of both study groups were compared. The uncertainty surrounding the cost-calculations was evaluated by means of standard bootstrap techniques. 27 Ultimately, the balance between costs and effects was compared for both strategies and incremental costs per therapy failure averted at 28 days were calculated. The uncertainty surrounding the incremental cost-effectiveness ratio was again evaluated by means of bootstrapping.

ELIGIBILITY:
Inclusion Criteria:

Adult patients (age 18 or above) with severe CAP admitted to general hospital wards were eligible for inclusion in the study. Pneumonia was defined as a new or progressive infiltrate on a chest X-ray plus at least two of the following criteria: cough, sputum production, rectal temperature > 38oC or < 36.1oC, auscultatory findings consistent with pneumonia, leucocytosis (>10.000/mm3, or >15% bands), C-reactive protein > 3 times the upper limit of normal, positive blood culture or positive culture of pleural fluid. 21 Severe pneumonia was defined as Fine class IV or V or fulfilling the ATS-criteria for severe community-acquired pneumonia

Exclusion Criteria:

Patients with cystic fibrosis, a history of colonization with Gram negative bacteria due to structural damage to the respiratory tract, malfunction of the digestive tract, life expectancy of less than 1 month due to underlying diseases, infections other than pneumonia needing antibiotic treatment, severe immunosuppression (neutropenia (<0,5 x 109 / l) or a CD4 count < 200 / mm3) and needing mechanical ventilation in an intensive care unit were excluded.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 2000-07; Study Completion 2004-03

PRIMARY OUTCOMES:
Clinical cure at day 28 of the study

SECONDARY OUTCOMES:
Costs for treatment both inside and outside the hospital
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Andy IM Hoepelman, Professor of Medicine, Principal Investigator — University Medical Center, Department of Internal Medicine and Infectious Diseases, Utrecht, The Netherlands
Locations (1):
- University Medical Center, Utrecht, Utrecht, Netherlands

REFERENCES:
- [Derived] Oosterheert JJ, Bonten MJ, Schneider MM, Buskens E, Lammers JW, Hustinx WM, Kramer MH, Prins JM, Slee PH, Kaasjager K, Hoepelman AI. Effectiveness of early switch from intravenous to oral antibiotics in severe community acquired pneumonia: multicentre randomised trial. BMJ. 2006 Dec 9;333(7580):1193. doi: 10.1136/bmj.38993.560984.BE. Epub 2006 Nov 7. PMID 17090560